CLINICAL TRIAL: NCT05434286
Title: Point-of-Care Echocardiography to Assess Impact of Dynamic Cardiac Function, Renal and Cardiac Biomarkers in Cirrhosis With Hepatorenal Syndrome-Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Department of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IM-2020-2145
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hepatorenal Syndrome; Cirrhosis, Liver; Acute-On-Chronic Liver Failure; AKI; Refractory Ascites
MeSH Terms: conditions — Hepatorenal Syndrome; Liver Cirrhosis; Acute-On-Chronic Liver Failure; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis/ACLF of any etiology: Cirrhosis with hepatorenal syndrome-acute kidney injury (HRS-AKI) as per International Ascites Club criteria.
  Interventions: Diagnostic Test: Echocardiographic assessment

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment — POC-Echocardiography to assess dynamic changes in cardiac output to assess therapeutic responses with albumin and terlipressin

SUMMARY:
Point-of-care echocardiography (POC-Echo) is used to determine left ventricular systolic and diastolic dysfunction (LVDD), inferior vena cava (IVC) dynamics and volume status in cirrhosis and Acute-on-chronic liver failure ACLF accurately.

We will assess IVC dynamics, LV systolic function [LV ejection fraction (EF) & cardiac output (CO)], and diastolic dysfunction (E/e', e' and E/A ratio) and urinary biomarkers (cystatin C and NGAL) in patients with cirrhosis and ACLF with hepatorenal syndrome-acute kidney injury (HRS-AKI).

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any Etiology
* Patient with acute kidney injury meeting HRS-AKI criteria

Exclusion Criteria:

* Hepatocellular carcinoma
* Patients with active variceal bleeding
* HIV or severe immunocompromised state
* Chronic kidney disease (CKD) on renal replacement therapy (RRT),
* Previous transjugular intra hepatic portosystemic shunt (TIPS)
* Porto-pulmonary hypertension,
* Coronary artery disease
* Congenital or valvular heart disease
* Prosthetic cardiac valves

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis of any etiology, aged between 18-65 years, with hepatorenal syndrome (HRS-AKI).
  Acute kidney injury (AKI) (increase in serum creatinine by 0.3 mg/dL in less than 48 hour or an increase in serum creatinine by 50% from a stable baseline reading within 3 months) has been proposed to characterize renal dysfunction in patients with cirrhosis, in which type 1 HRS would be reclassified as HRS-AKI.
  Stage 1 AKI would be classified as an increase in serum creatinine level by 0.3 mg/dL or a 50% increase, whereas stages 2 and 3 AKI would be a doubling and tripling, respectively, of serum creatinine levels.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measurement by echocardiography | Day 0, Day 2, Day 7.
  Echocardiographic assessment of cardiac output in L/min will be recorded at least 3 time points, day 0 and 48 hours after enrollment.
  The cardiac output at 7 days after enrollment will also be documented. he Doppler velocity time integral (VTI) method in estimating stroke volume and cardiac output correlates well with results of concurrent thermodilution cardiac output determinations in patients without significant left-sided valvular regurgitation.
  Cardiac output(CO), Stroke volume (SV), Heart rate (HR)
  CO = [SV * HR]/ 1000
IVC size and collapsibility changes | Day 0.
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
IVC size and collapsibility changes | Day 2
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
IVC size and collapsibility changes | Day 7.
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
Number of patients with Complete Response in HRS-AKI | Day 7
  Complete response is defined as a reversal in AKI with a final serum Creatinine (sCr) value of ≤ 0.3 mg/dL of the baseline.
Number of patients with Partial Response in HRS-AKI | Day 7
  Partial response is defined as regression in the stage of AKI with a final sCr > 0.3 mg/dL above the baseline.
Number of patients with Non-Response in HRS-AKI | Day 7
  Non-responder is defined if the sCr did not decrease or increased from the baseline.

SECONDARY OUTCOMES:
Change in Cystatin C and Neutrophil gelatinase associated lipocalin (NGAL) level | Day 0 and Day 7
Change in NT Pro brain natriuretic peptide (BNP) level | Day 0 and Day 7
Change in plasma renin activity level | Day 0 and Day 7
Change in Galectin-3 level | Day 0 and Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Adebayo D, Neong SF, Wong F. Refractory Ascites in Liver Cirrhosis. Am J Gastroenterol. 2019 Jan;114(1):40-47. doi: 10.1038/s41395-018-0185-6. PMID 29973706
- [Derived] Premkumar M, Kajal K, Reddy KR, Izzy M, Kulkarni AV, Duseja AK, Sihag KB, Divyaveer S, Gupta A, Taneja S, De A, Verma N, Rathi S, Bhujade H, Chaluvashetty SB, Roy A, Kumar V, Siddhartha V, Singh V, Bahl A. Evaluation of terlipressin-related patient outcomes in hepatorenal syndrome-acute kidney injury using point-of-care echocardiography. Hepatology. 2024 May 1;79(5):1048-1064. doi: 10.1097/HEP.0000000000000691. Epub 2023 Nov 16. PMID 37976391